CLINICAL TRIAL: NCT00703937
Title: A Multi-center, Randomized, Controlled Study to Investigate the Safety and Tolerability of Intravenous Ferric Carboxymaltose (FCM) vs. Standard Medical Care in Treating Iron Deficiency Anemia
Brief Title: Safety and Tolerability of Ferric Carboxymaltose (FCM) Versus Standard of Care in Treating Iron Deficiency Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT08019
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose; Clinical Trials Data Monitoring Committees

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferric Carboxymaltose (FCM) (Experimental): 750 mg of iron as undiluted FCM (15 mg/kg up to a maximum of 750 mg) at 100 mg per minute weekly until the calculated iron deficit dose has been administered (to a maximum cumulative dose of 2,250 mg).
  Interventions: Drug: Ferric Carboxymaltose (FCM)
- Standard Medical Care (SMC) for the treatment of IDA (Active Comparator): SMC as determined by the Investigator for the treatment of iron deficiency anemia (IDA).
  Interventions: Drug: Standard Medical Care (SMC) for the treatment of IDA

INTERVENTIONS:
Drug: Ferric Carboxymaltose (FCM)
  Arms: Ferric Carboxymaltose (FCM)
Drug: Standard Medical Care (SMC) for the treatment of IDA
  Arms: Standard Medical Care (SMC) for the treatment of IDA

SUMMARY:
The objective of this study is to evaluate the safety of FCM in patients with anemia who are not dialysis dependent.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age and able to give informed consent
* Iron deficiency is the primary etiology of anemia
* Screening Visit central laboratory Hemoglobin (Hgb) ≤ 11g/dL
* Screening Visit ferritin ≤ 100ng/mL or ≤ 300 ng/mL when TSAT was ≤ 30%

Exclusion Criteria:

* Previous participation in a FCM trial
* Known hypersensitivity reaction to FCM
* Requires dialysis for treatment of chronic kidney disease
* Current anemia not attributed to iron deficiency
* Received IV iron, RBC transfusion(s), or antibiotics 10 days prior and during the screening phase
* Anticipated need for surgery
* AST or ALT greater than 1.5 times the upper limit of normal
* Received an investigational drug within 30 days of screening
* Pregnant or sexually-active females who are not willing to use an effective form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals, Norristown, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals and medical clinics
Pre-assignment Details: 5 subjects randomized into the trial were discontinued prior to dosing.
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care (SMC) for the Treatment of IDA
Started | 343 | 360
Completed | 278 | 267
Not Completed | 65 | 93

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care (SMC) for the Treatment of IDA | Total
Number analyzed (Participants) | 343 | 360 | 703
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 3 | 4
  Between 18 and 65 years | 267 | 287 | 554
  >=65 years | 75 | 70 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (18.48) | 47.7 (17.62) | 48.5 (18.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 292 | 318 | 610
  Male | 51 | 42 | 93
Region of Enrollment [Number; unit: participants]
  United States | 343 | 360 | 703

OUTCOME MEASURES:

1. Primary Outcome: Safety, as Defined by the Occurence of Serious Adverse Events (SAE's), of FCM Compared to SMC
Description: Safety, as defined by the occurence of serious adverse events (SAE's), of FCM compared to SMC in the treatment of IDA in subjects who were not dialysis dependent
Time Frame: First administration of FCM, or Day 0 for SMC subjects, through end of study (Day 42) or 28 days after the last dose of study drug (FCM or SMC) whichever was longer
Measure: Number; unit: participants
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care (SMC) for the Treatment of IDA
Number analyzed (Participants) | 343 | 360
participants | 17 | 11

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ferric Carboxymaltose (FCM) | Standard Medical Care (SMC) for the Treatment of IDA
Serious Adverse Events (participants affected / at risk) | 17/343 | 11/360
Other Adverse Events (participants affected / at risk) | 41/343 | 71/360
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=343) | Standard Medical Care (SMC) for the Treatment of IDA (N=360)
Anemia (Blood and lymphatic system disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cartoid artery stenosis (Nervous system disorders) | 1 | 0
Facial palsy (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal infarct (Renal and urinary disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 2
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=343) | Standard Medical Care (SMC) for the Treatment of IDA (N=360)
Constipation (Gastrointestinal disorders) | 12 | 26
Nausea (Gastrointestinal disorders) | 14 | 27
Headache (Nervous system disorders) | 16 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less